CLINICAL TRIAL: NCT02383186
Title: Dermal Suturing Only Versus Layered Cutaneous Closure: A Randomized Split Wound Comparative Effectiveness Trial
Brief Title: Dermal Suturing Only Versus Layered Cutaneous Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 614521
Record Dates: First submitted 2014-11-10; First posted 2015-03-09 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Wound Closure Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dermal Suturing Only Wound Closure (Active Comparator): The side assigned to dermal suturing only will be closed with a single layer of deep absorbable sutures. The method will be buried vertical mattress or set-back suturing at the surgeons discretion.
  Interventions: Procedure: Dermal Suturing Only Wound Closure; Procedure: Layered Cutaneous Wound Closure
- Layered Cutaneous Wound Closure (Active Comparator): The side assigned to layered closure is closed with 5-0 fast acting gut.
  Interventions: Procedure: Dermal Suturing Only Wound Closure; Procedure: Layered Cutaneous Wound Closure

INTERVENTIONS:
Procedure: Dermal Suturing Only Wound Closure — The side assigned to dermal suturing only will be closed with a single layer of deep absorbable sutures. The method will be buried vertical mattress or set-back suturing at the surgeons discretion.
Procedure: Layered Cutaneous Wound Closure — The side assigned to layered closure is closed with 5-0 fast acting gut.

SUMMARY:
The purpose of this study is to determine whether a single layer dermally sutured wound results in superior outcomes to a layered closure.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a single layer dermally sutured wound results in superior outcomes to a layered closure. Our aims are to compare outcomes using a split wound model, where half the wound is sutured with one technique and the other half is sutured with the other. This will be measured via the physician observer scar assessment scale, a validated scar instrument and via wound width. Our hypothesis is that wounds with a single layer closure will result in cosmetically superior wound outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure with predicted linear closure
* Willing to return for follow up visits

Exclusion Criteria:

* Mentally handicapped
* Incarceration
* Pregnant Women
* Wounds with predicted closure length less than 3 cm
* Wounds unable to be fully closed via primary closure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05-28 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Assessment of Scar on the Patient and Observer Scar Assessment Scale at 3 Months | 3 months
  After surgical procedure, half of the subject's wound will be closed by single layer suturing, while the other half is closed by layered cutaneous closure. After 3 months, subjects will return to clinic for evaluation of the cosmesis of both types of closure techniques.
Assessment of Scar on the Patient and Observer Scar Assessment Scale at 12 Months | 12 months
  After surgical procedure, half of the subject's wound will be closed by single layer suturing, while the other half is closed by layered cutaneous closure. After 12 months, subjects will return to clinic for evaluation of the cosmesis of both types of closure techniques.

SECONDARY OUTCOMES:
Measurement of Scar Width | 3 months and 12 months
  The width of the scar will be measured 1 centimeter from the midline on both sides. There is no defined width that is considered satisfactory or not satisfactory. The measurements will be compared between subjects.
Assessment of Complications | 3 months and 12 months
  Noting the presence or absence of bleeding, dehiscence, infection or spitting sutures.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, M.D., Principal Investigator — University of California, Davis

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical